CLINICAL TRIAL: NCT01300325
Title: Effectiveness of Nebulized Hypertonic Saline and Epinephrine in Hospitalized Infants With Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Michele Miraglia, Dipartimento di Pediatria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENHS
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-01

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis, 3% Hypertonic Saline Solution
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.9% saline (Placebo Comparator): patients receive every 6 hours the nebulized 0.9% saline (placebo comparator) (group I) or the 3% HS (group II) in addition to aerosolized epinephrine (1.5 mg) and to the conventional treatment (oxygen, fluids).
  Interventions: Other: 3% hypertonic saline solution
- 3% hypertonic saline (No Intervention): Patients receive every 6 hours the nebulized 0.9% saline (Placebo comparator) (group I) or the 3% hypertonic saline solution group II) in addition to aerosolized epinephrine (1.5 mg) and to the conventional treatment (oxygen, fluids).

INTERVENTIONS:
Other: 3% hypertonic saline solution — Patients receive every 6 hours the nebulized 0.9% saline (Placebo comparator) (group I) or the 3% hypertonic saline solution group II) in addition to aerosolized epinephrine (1.5 mg) and to the conventional treatment (oxygen, fluids).
  Arms: 0.9% saline

SUMMARY:
Acute bronchiolitis is the main cause for respiratory illness that requires hospitalization in children younger than 2 years. In the United States it has been shown that the burden of the disease is considerable, having an annual cost of more than $ 500 million and being responsible for the 17% of all infant hospitalizations . Aim of the present study was to verify the effects of nebulized 3% saline solution in comparison to normal saline in addiction to epinephrine in a large population of RSV positive cases of bronchiolitis; all patients presented a disease as much as severe to require hospitalization.The main study endpoints were the length of stay in hospital and the clinical response.

DETAILED DESCRIPTION:
Among 136 patients assessed within 12 hours for entry into the study, 109 (69 males) accepted to participate, gave an informed consent and were randomly assigned either to receive every 6 hours the nebulized 0.9% saline (NS) (group I) or the 3% HS (group II) in addition to aerosolized epinephrine (1.5 mg) and to the conventional treatment (oxygen, fluids). Patients were randomized to receive different saline treatments using a computer-based randomization program. Study solutions, prepared by the local hospital pharmacy, were blinded to participants and investigators. Each treatment was delivered by a nebulizer with continuous flow of oxygen at 6 L/min through a tight-fitting facemask.

The main study endpoints were the length of stay (LOS) in hospital and the clinical response. LOS in hospital was defined as the time between study entry (within 12 hours of admission to the hospital) and the time at which the infant was discharged on the basis of the clinical grounds by the attending physician. Clinical response was determined using daily CSS evaluation; furthermore, the CSS was evaluated every day before and 30 minutes after nebulisation.

ELIGIBILITY:
Inclusion Criteria:

* children aged less than 2 years old
* clinical diagnosis of bronchiolitis

Exclusion Criteria:

* cardiac or pulmonary diseases
* premature birth < 36 weeks of gestational age
* previous diagnosis of asthma
* an initial oxygen saturation of 85%

Ages: 30 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
time of hospitalization | six days
  length of stay

SECONDARY OUTCOMES:
Clinical response before and 30 minutes after nebulisation by score | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michele Miraglia, MD, Study Director — Pediatric Department
Locations (1):
- Azienda Sanitaria Locale Napoli 2 Nord, Pozzuoli, Napoli, Italy